CLINICAL TRIAL: NCT06652087
Title: The Effect of Correction of Bacterial Overgrowth Syndrome in the Small Intestine on Cardiac Function in Patients with Heart Failure with Preserved Ejection Fraction
Brief Title: Rifaximin and Cardiac Function in Patients with Heart Failure with Preserved Ejection Fraction
Acronym: SIBO-HFpEF
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: I.M. Sechenov First Moscow State Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: VI27478
Record Dates: First submitted 2024-09-09; First posted 2024-10-22 (Actual); Last update posted 2024-10-22 (Actual); Status verified 2024-09

CONDITIONS: Bacterial Overgrowth Syndrome Small Bowel; Heart Failure with Preserved Ejection Fraction
Keywords: Chronic heart failure with preserved ejection fraction; Diastolic dysfunction; Overweight; Obesity; The gut-heart axis; Small intestinal bacterial overgrowth syndrome
MeSH Terms: conditions — Overweight; Obesity | interventions — Rifaximin

STUDY DESIGN:
Intervention Model Description: The participants are divided into two parallel groups for the duration of the study. Forty patients with HFRS with a body mass index of more than 25 kg/m2 and a positive SIBO test will be randomly assigned in a 1:1 ratio to the experimental (rifaximin) and control groups. All patients will also receive standard HF treatment (diuretics, including an aldosterone antagonist; a sodium-glucose cotransporter-2 inhibitor).
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- intervention group (Experimental): Patients of the experimental group will receive standart therapy HFpEF and rifaximin (Alfa Normix®, Alfa Wassermann S.P.A., Italy, registration number LS-001993, 08/31/2010) at a dose of 200 mg 3 times a day for 7 days.
  Interventions: Drug: Rifaximin; Other: Standard HFpEF treatment
- control group (Active Comparator): Patients of the control group will receive standart therapy HFpEF Without Rifaximin
  Interventions: Other: Standard HFpEF treatment

INTERVENTIONS:
Drug: Rifaximin — Rifaximin (Alfa Normix®, Alfa Wassermann S.P.A., Italy, registration number LS-001993, 08/31/2010) in standard doses of 200 mg 3 times a day for 7 days
  Other Names: Alfa Normix®
  Arms: intervention group
Other: Standard HFpEF treatment — diuretic, including an aldosterone antagonist; sodium-glucose cotransporter-2 inhibitor

SUMMARY:
Single-center, double-blind, randomized, controlled intervention study of the effect of correction of bacterial overgrowth syndrome in the small intestine (SIBO) on cardiac function in patients with heart failure with preserved ejection fraction (HFpEF) (SIBO-HFpEF). The aim of the study is to evaluate the efficacy and safety of rifaximin in patients with HFpEF and SIBO.

DETAILED DESCRIPTION:
The proportion of patients with obvious symptoms of chronic heart failure with preserved ejection fraction (HFpEF) is more than 50%, and mortality is comparable to that of patients with low ejection fraction. The lack of evidence regarding therapeutic possibilities for improving the prognosis leads to the search for new treatment regimens. Systemic low-grade inflammation is recognized as the fundamental pathophysiological mechanism of HFpEF. On the one hand, it is caused by obesity, which is the background for the comorbidity of these patients. On the other hand, chronic sluggish systemic inflammation in combination with changes in the composition and metabolic activity of the gut microbiota, dysfunction of the intestinal barrier explains the role of the gut-heart axis in the pathogenesis of HFpEF. There is evidence that small intestinal bacterial overgrowth syndrome (SIBO) is an independent risk factor for re-hospitalization and cardiovascular death among all patients with heart failure. SIBO and its correction in patients with HFpEF have not been sufficiently studied.

Forty patients with HFpEF with a body mass index of more than 25 kg/m2 and a positive SIBO test will be randomly assigned in a ratio of 1:1 to the experimental (rifaximin) and control groups. To detect SIBO, a hydrogen breathing test with lactulose (Duphalac®, Abbott Biologicals B.V., the Netherlands, registration number N011717/02 dated 02/04/2010) will be performed on a medical device "Respiratory hydrogen Gastro+ Gastrolyzer®(EC60) with accessories" (Bedfont Scientific Ltd., Great Britain, registration number 2010/06253 dated 09/17/2020). For 2 hours, every 15 minutes, the patient will be asked to take a deep breath, hold his breath for 10-15 seconds and exhale into a special device for measuring the concentration of hydrogen in the exhaled air. Interpretation of a positive result (threshold of increase from the zero point): ≥20 ppm. Patients in the experimental group (SIBO positive test) will be prescribed rifaximin (Alfa Normix®, Alfa Wassermann S.P.A., Italy, registration number LS-001993, 08/31/2010) in standard doses of 200 mg 3 times a day for 7 days. Patients from the control group (positive SIBO test) will not receive rifaximin. All patients will also receive standard HFpEF treatment (diuretic, including an aldosterone antagonist; sodium-glucose cotransporter-2 inhibitor). Patients will be blinded. A control breath test with lactulose will be performed after completion of rifaximin intake and one month after discharge from the hospital. Markers of systemic inflammation in the blood (levels of C-reactive protein, fibrinogen and ferritin) and parameters of diastolic dysfunction (transthoracic echocardiography) will also be evaluated. After the end of the study, an analysis of the effect of adding rifaximin to the standard treatment of CHF compared with the control group will be carried out.Patients from the control group (with a positive SIBO test result) will not receive rifaximin. All patients will also receive standard treatment for HFRS (diuretics, including an aldosterone antagonist; a sodium-glucose cotransporter-2 inhibitor). Patients will be blinded. A control breath test with lactulose will be performed after completion of rifaximin and one month after discharge from the hospital. Markers of systemic inflammation in the blood (levels of C-reactive protein, fibrinogen and ferritin) and parameters of diastolic dysfunction (transthoracic echocardiography) will also be evaluated. After the end of the study, the effect of adding rifaximin to the standard treatment of CHF will be analyzed compared with the control group. Researchers suggest that rifaximin reduces the level of markers of systemic inflammation, reduces the severity of diastolic dysfunction, is effective in SIBR in patients with HF and BMI≥25 kg/m2, improves their quality of life and prognosis. Patients from the control group (with a positive SIBO test result) will not receive rifaximin. All patients will also receive standard treatment for HFRS (diuretics, including an aldosterone antagonist; a sodium-glucose cotransporter-2 inhibitor). Patients will be blinded. A control breath test with lactulose will be performed after completion of rifaximin and one month after discharge from the hospital. Markers of systemic inflammation in the blood (levels of C-reactive protein, fibrinogen and ferritin) and parameters of diastolic dysfunction (transthoracic echocardiography) will also be evaluated. After the end of the study, the effect of adding rifaximin to the standard treatment of CHF will be analyzed compared with the control group. Researchers suggest that rifaximin reduces the level of markers of systemic inflammation, reduces the severity of diastolic dysfunction, is effective in SIBR in patients with HF and BMI≥25 kg/m2, improves their quality of life and prognosis.

ELIGIBILITY:
Inclusion Criteria:

1. availability of written informed consent of the patient to participate in the study
2. adult aged ≥18≤80 years' old
3. body mass index ≥25 kg/m2
4. diagnosed with HFpEF: 1) symptoms and/or signs of heart failure; 2) left ventricular ejection fraction ≥50%; 3) increased levels of natriuretic peptides (NTproBNP≥125 pg/mL); 4) at least one additional criterion: relevant structural heart disease (hypertrophy of the left ventricle (LVH) and/or enlargement of the left atrium (LAE) or diastolic dysfunction

Exclusion Criteria:

1. refusal of the patient from further participation in the study
2. identification of any disease or condition specified in the criteria for non-inclusion and the development of a severe pathological condition in which patient monitoring becomes poorly implemented and the presence of which may make it difficult to interpret the data (gastrointestinal bleeding, myocardial infarction, etc.)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-09-02 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
Changing the functional class (FC) of chronic heart failure (CHF) | Day 1, day 10, day 40
  The 6-Minute Walk Distance (6-MVD) The test will be conducted according to the standard procedure in a marked corridor (length 50 meters) in the morning. Each patient needs to walk the maximum possible distance along the corridor at an acceptably fast pace in 6 minutes. Interpretation of the results in relation to the classification of the New York Heart Association Classification: 426- 550 m corresponds to FC I, 301-425 m corresponds to FC II, 151-300 m corresponds to FC III, less than 150 m corresponds to FC IV.
Change in clinical condition | Day 1, day 40
  Clinical Condition Assessment Scale (CCAS) (in the modification of Mareev V.Yu., 2000) This scale includes 10 points (depending on the result, each answer is assigned a certain number of points, which are summed up): shortness of breath (0 - no, 1 - under load, 2 - at rest), weight change over the last week (0 - no, 1 - increased), complaints of irregular heartbeat (0 - no, 1 - there is), the patient's position in bed (0 - horizontally, 1 - with raised headboard (+2 pillows), 2 - plus wakes up from suffocation, 3 - sitting), swollen cervical veins (0 - no, 1 - lying down, 2 - standing), wheezing in the lungs (0 - no, 1 - lower parts (up to 1/3), 2 - up to the shoulder blades (up to 2/3), 3 - over the entire surface of the lungs), the presence of a gallop rhythm (0 - no, 1 - there is), liver (0 - not enlarged, 1 - up to 5 cm, 2 - more than 5 cm), edema (0 - no, 1 - pastosity, 2 - edema, 3 - anasarca), the level of systolic blood pressure (0 - >120, 1 - 100-200, 2 - <100 mmHg). Summary

SECONDARY OUTCOMES:
Changes in the level of C-reactive protein in blood serum | Day 1, day 40
  Venous blood will be taken on an empty stomach at 7-9 am without any special preparation
Changes in serum fibrinogen levels | Day 1, day 40
  Venous blood will be taken on an empty stomach at 7-9 am without any special preparation
Changes in serum ferritin levels | Day 1, day 40
  Venous blood will be taken on an empty stomach at 7-9 am without any special preparation
Change in the presence of the small intestinal bacterial overgrowth | Day 2, day 10, day 40
  Hydrogen breathing test with lactulose on Gastro+ Gastrolyzer (EC60) (Bedfont Scientific Ltd., Great Britain, registration number 2010/06253 dated 09/17/2020) in accordance with the North American consensus: the presence of excessive bacterial growth in the small intestine is considered when the hydrogen content in the breath is increased by at least 20 ppm above the initial value for 90 minutes after taking 10 ml of lactulose dissolved in 200 ml of water
Change in the maximum volume of the left atrium indexed to the body surface area | Day 1, day 40
  Transthoracic echocardiography (GE VIVID E95, "GE Vingmed Ultrasound AS", Norway, registration certificate 2016/3871 dated 10/17/2022) will be performed at 10-12 am without any special preparation
Change in the ratio of the maximum rates of early diastolic transmittal blood flow (E) and diastolic elevation of the base of the left ventricle in the early diastole (e') Е/e' | Day 1, day 40
  Transthoracic echocardiography (GE VIVID E95, "GE Vingmed Ultrasound AS", Norway, registration certificate 2016/3871 dated 10/17/2022) will be performed at 10-12 am without any special preparation
Change in tricuspid regurgitation | Day 1, day 40
  Transthoracic echocardiography (GE VIVID E95, "GE Vingmed Ultrasound AS", Norway, registration certificate 2016/3871 dated 10/17/2022) will be performed at 10-12 am without any special preparation

CONTACTS AND LOCATIONS:
Overall Officials: Vladimir Ivashkin, Principal Investigator — I.M. Sechenov First Moscow State Medical University (Sechenov University)
Locations (1):
- Moscow, Moscow, Russia

IPD SHARING:
Plan to Share IPD: No
The disclosure of data is not allowed by the Local Ethics Committee of the I.M. Sechenov First Moscow State Medical University (Sechenov University).